CLINICAL TRIAL: NCT02415166
Title: Influenza Challenge in Mood Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LIBR # 2015-001-00
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: MAJOR DEPRESSIVE DISORDER
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- VACCINE MDD (Experimental): SEASONAL INFLUENZA VACCINE (0.5ML) DELIVERED I.M.
  Interventions: Biological: INFLUENZA VACCINE
- PLACEBO MDD (Placebo Comparator): SALINE (0.5ML) DELIVERED I.M.
  Interventions: Other: NaCl-saline placebo
- VACCINE HC (Experimental): SEASONAL INFLUENZA VACCINE (0.5ML) DELIVERED I.M.
  Interventions: Biological: INFLUENZA VACCINE
- PLACEBO HC (Placebo Comparator): SALINE (0.5ML) DELIVERED I.M.
  Interventions: Other: NaCl-saline placebo

INTERVENTIONS:
Biological: INFLUENZA VACCINE — THE PURPOSE OF THE STUDY IS TO EVALUATE THE EFFICACY OF THE SEASONAL INFLUENZA VACCINE IN PEOPLE WITH MAJOR DEPRESSIVE DISORDER
  Arms: VACCINE HC; VACCINE MDD
Other: NaCl-saline placebo — placebo
  Arms: PLACEBO HC; PLACEBO MDD

SUMMARY:
The aim of this project is to evaluate the efficacy of the influenza vaccine in individuals with major depressive disorder (MDD) as well as to elucidate the nature of the immunological abnormalities in MDD using a quasi-experimental design. Specifically, the investigators plan to induce transient, mild inflammation in medically-healthy study participants using the influenza vaccine. Initially the investigators will conduct a pilot project with up to 20 individuals in order to evaluate the time-point at which the peak inflammatory response to the vaccine occurs. Subjects will receive the seasonal influenza vaccine and provide blood samples 4 hours, 2 days, and 30 days post vaccination. Subsequent to the pilot study, both depressed and psychiatrically-healthy participants will be randomized in a parallel group, double-blind design so that they receive either influenza vaccine (seasonal vaccine) or saline (i.m). At baseline, subjects will provide a blood sample, complete a number of rating scales to measure mood and fatigue, and may complete approximately one hour of MRI scanning with or without simultaneous EEG recording. Two-days post vaccination, they will provide a second blood sample, complete more clinical ratings and may complete another identical MRI session with or without simultaneous EEG. Four weeks later, participants will be asked to return to provide a third blood sample and complete additional clinical ratings. The blood samples will be used to measure both innate and adaptive immune function and may be used to correlate the vaccine-induced immunological changes to neurophysiological changes in the brain measured by MRI and/or EEG.

DETAILED DESCRIPTION:
Psychological stress has been shown to impair the efficacy of the influenza vaccine, particularly in older individuals (> 60 years). However, the effect of depression (as opposed to stress per se) on vaccine response has not been measured, especially in younger people. One possible cause of this putative impaired vaccine response is suppression of the immune system in a subgroup of individuals with depression. Major depressive disorder (MDD) has been associated with a decline in total numbers of circulating B-cells, T-cells, and natural killer cells (NKC), a reduction in the proliferative responses of NKC and T-cells in vitro that is ameliorated by administration of selective serotonin reuptake inhibitors (SSRIs), increased susceptibility to various viral infections, and a decline in the efficacy of the herpes zoster vaccine in the elderly (1, 2). On the other hand, MDD appears also to be characterized by immunological abnormalities that manifest both as low-grade inflammation, including over-activity of the innate immune system (3). Whether inflammation and immune suppression are two different manifestations of the same underlying abnormality (unitary model) or whether inflammation and immune suppression are distinct phenomena occurring in different MDD subtypes (independent model) is not known.

MDD is also characterized by neurophysiological abnormalities of striatal, cortical midline, and limbic brain structures that regulate hormonal, autonomic, and emotional responses to reward and stress (4-6). Yet, it remains unclear how immune function relates to these depression-associated functional neuroimaging abnormalities. Studies of healthy volunteers (HCs) administered endotoxin or the typhoid vaccine have reported inflammation-associated increases in negative affect along with neurophysiological changes in brain regions comprising the affective and reward circuitry (7-8). However, because these studies were limited to HCs, it is possible that the observed inflammation-induced neurophysiological changes were adaptive and therefore not applicable to MDD populations. That is, it remains unclear whether any experimentally-induced immune abnormalities in MDD are correlated and therefore potentially causally-related to the neuroimaging abnormalities observed in MDD.

In order to address these questions, we use a parallel group, placebo-controlled influenza vaccine challenge to induce transient inflammation that peaks 2-days post vaccination in MDD subjects and HCs. Subjects may complete a pre-and-post vaccination MRI scan, the latter during the peak inflammatory response.

Aim 1: To examine whether influenza vaccine effectiveness is compromised in a young-to-middle-aged sample (18-55 years of age) of individuals with MDD.

Hypothesis 1.1. Compared with HCs (n=40), individuals with MDD (n=40) will display reduced vaccine titers and reduced influenza virus-induced CD4+ memory T-cell proliferation four weeks post vaccination (T2).

Hypothesis 1.2. A greater number of MDD subjects than HCs will fail to show a four-fold increase in antibody titer, the conventional standard for determining a clinically significant response to a viral vaccine.

Aim 2: To test the competing models of immune dysfunction in MDD.

Hypothesis 2.1. At T0 and T1, stimulated and unstimulated monocytes from MDD subjects will show increased interleukin 6 (IL-6) and tumor necrosis factor (TNF) production compared with HCs. The effect will be most salient at T1 in individuals receiving vaccine.

Hypothesis 2.2. Consistent with the unitary model, monocyte IL-6 and/or TNF production at T0 and T1 will be inversely correlated with antibody titers at T2 in the MDD group.

Aim 3: To test for neurophysiological differences between MDD patients and HCs in resting state cerebral blood flow (with arterial spin labeling), resting EEG activity, and BOLD response to monetary rewards and interoceptive stimuli (with fMRI) at T0 and T1, and to correlate depression-associated perfusion, EEG activity, reward response, and interoceptive function with immune function at T0 and T1.

Hypothesis 3.1: Compared with HCs, the MDD subjects will display reduced perfusion of the subgenual anterior cingulate cortex (sgACC) and/or pregenual ACC (pgACC), hemispheric asymmetry in the alpha (8-13 Hz) power band (left prefrontal cortex hypoactivation), as well as reduced hemodynamic response to anticipatory reward in the ventral striatum. These differences will be most salient at T1 in the MDD group receiving vaccine versus the HCs receiving vaccine.

Hypothesis 3.2: The functional imaging abnormalities in the MDD group at T0 and/or T1 will be correlated with the abnormalities in monocyte activation in the MDD group at T0 and/or T1.

ELIGIBILITY:
Inclusion Criteria:

Major Depressive Disorder Patient Group - Currently Depressed: Subjects will have met Diagnostic and Statistical Manual of the American Psychiatric Association (DSM-V) criteria for primary MDD in a current major depressive episode and current Hamilton Depression Rating Scale (HAM-D) or Montgomery Asberg Depression Rating Scale (MADRS) score in the mild-to-severely depressed range and will have been deemed to be medically stable by a physician listed on this protocol. Subjects who do not wish to receive treatment with psychotropic medication in the future and have not taken psychotropic medication for at least 3 weeks will be included in the study.

Healthy Comparison Group: Subjects will be selected who have not met criteria for any Axis I psychiatric disorder, have no known first-degree relatives with mood or anxiety disorders, and have a current score on the HAM-D or MADRS in the non-depressed range.

Exclusion Criteria:

Inability to provide informed consent, pregnant or nursing women, known hypersensitivity to vaccines, age of onset of MDD > 40 years, metal implants or other factors that would preclude MRI scanning, serious risk of suicide, delusions or hallucinations, medical or neurological illnesses (such as diabetes, autoimmune disorders or inflammatory bowel disease) that affect brain structure, function or immune measurements, previous head injury with loss of consciousness, abuse of drugs or alcohol within the previous year or a lifetime history of substance dependence, treatment with medications that impact immune function (e.g. prednisone), HIV or other chronic infection, a recent acute illness (e.g. influenza), receipt of a vaccine within 3 months of commencing the study. Subjects whose first major depressive episodes arose temporally after other major medical or psychiatric conditions will also be excluded, since their functional imaging results generally differ from those reported in primary MDD.

Subjects will be asked not to take any over-the-counter non-steroidal anti-inflammatory drugs or drink alcohol for 48 hr. before each study day. The use of oral contraceptives and menstrual phase or status are not exclusion criteria but this information will be recorded. The same exclusion criteria apply to healthy controls with the added criterion that first-degree relatives should be free of major psychiatric illness as assessed with the Family Interview for Genetic Studies (FIGS).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Savitz, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brian Research, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Irwin MR, Miller AH. Depressive disorders and immunity: 20 years of progress and discovery. Brain Behav Immun. 2007 May;21(4):374-83. doi: 10.1016/j.bbi.2007.01.010. Epub 2007 Mar 13. PMID 17360153
- [Background] Blume J, Douglas SD, Evans DL. Immune suppression and immune activation in depression. Brain Behav Immun. 2011 Feb;25(2):221-9. doi: 10.1016/j.bbi.2010.10.008. Epub 2010 Oct 16. PMID 20955778
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Price JL, Drevets WC. Neurocircuitry of mood disorders. Neuropsychopharmacology. 2010 Jan;35(1):192-216. doi: 10.1038/npp.2009.104. PMID 19693001
- [Background] Robinson OJ, Cools R, Carlisi CO, Sahakian BJ, Drevets WC. Ventral striatum response during reward and punishment reversal learning in unmedicated major depressive disorder. Am J Psychiatry. 2012 Feb;169(2):152-9. doi: 10.1176/appi.ajp.2011.11010137. PMID 22420038
- [Background] Savitz J, Drevets WC. Bipolar and major depressive disorder: neuroimaging the developmental-degenerative divide. Neurosci Biobehav Rev. 2009 May;33(5):699-771. doi: 10.1016/j.neubiorev.2009.01.004. Epub 2009 Jan 21. PMID 19428491
- [Background] Eisenberger NI, Berkman ET, Inagaki TK, Rameson LT, Mashal NM, Irwin MR. Inflammation-induced anhedonia: endotoxin reduces ventral striatum responses to reward. Biol Psychiatry. 2010 Oct 15;68(8):748-54. doi: 10.1016/j.biopsych.2010.06.010. Epub 2010 Aug 16. PMID 20719303
- [Background] Harrison NA, Brydon L, Walker C, Gray MA, Steptoe A, Critchley HD. Inflammation causes mood changes through alterations in subgenual cingulate activity and mesolimbic connectivity. Biol Psychiatry. 2009 Sep 1;66(5):407-14. doi: 10.1016/j.biopsych.2009.03.015. Epub 2009 May 7. PMID 19423079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated after the recruitment of six participants
Period: Overall Study
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Started | 6 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC | Total
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 6 |  |  |  | 6
  >=65 years | 0 |  |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (6) |  |  |  | 35 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  |  | 4
  Male | 2 |  |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 |  |  |  | 6

OUTCOME MEASURES:

1. Primary Outcome: THE TITER OF INFLUENZA ANTIBODIES
Description: Outcome data were not collected.
  This was a failed study as all participants, including those who were putatively vaccine-naive had antibodies to influenza at baseline and therefore the original hypothesis could not be tested. The study was terminated.
Time Frame: ONE MONTH
Population: Unmedicated outpatients with major depressive disorder. Outcome data not collected.
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: THE INFLUENZA VIRUS-INDUCED PROLIFERATION OF CD4+ MEMORY T-CELLS
Description: Data not collected.
Time Frame: ONE MONTH
Population: Unmedicated participants with major depressive disorder. Data were not collected.
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: IL-6 AND TNF PRODUCTION BY STIMULATED AND UNSTIMULATED MONOCYTE CELLS
Time Frame: 2 DAYS
Population: Data not analyzed
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: DIFFERENCES IN RESTING STATE CEREBRAL BLOOD FLOW BETWEEN MDD AND HC GROUPS
Time Frame: 2 DAYS
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: DIAGNOSTIC GROUP DIFFERENCES IN THE BOLD RESPONSE (Using fMRI) TO MONETARY REWARDS IN THE VENTRAL STRIATUM
Time Frame: 2 DAYS
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | VACCINE MDD | PLACEBO MDD | VACCINE HC | PLACEBO HC
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a failed study as all participants, including those who were putatively vaccine-naive had antibodies to influenza at baseline and therefore the original hypothesis could not be tests. The study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes